CLINICAL TRIAL: NCT03317782
Title: Evaluation of NoL Index Variations After a Painful Stimulus Before and After a Stellate Ganglion Block in Patients With Upper Extremity Complex Regional Pain Syndrome: a Pilot Study
Brief Title: NoL Index Variations Before and After a Stellate Ganglion Block
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, Dr, Maisonneuve-Rosemont Hospital
Other Study IDs: 2017-1072
Record Dates: First submitted 2017-10-14; First posted 2017-10-23 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: NoL index — The NoL/PMD-200 (Medasense Biometrics Ltd, Ramat Yishai, Israel) is a multi-parameter index (0-100) that incorporates heart rate, heart rate variability (0.15-0.4 Hz band power), plethysmograph wave amplitude, skin conductance level, number of skin conductance fluctuations (NSCF), and their time derivatives9 using a non-linear regression technique. A higher index indicates higher nociception, and an index <20 indicates adequate analgesia.

SUMMARY:
To evaluate and compare the NoL index variations after a painful physiotherapy exercise in patients with upper limb CRPS, before and after a stellate ganglion block.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of upper limb CRPS according to the Budapest criteria12, for more than 6 months;
* Significant pain relief from stellate ganglion block;
* Undergoing physical therapy;
* 18 years and older.

Exclusion Criteria:

* Patients taking beta blockers

  * Bilateral/generalized CRPS
  * Patients needing sedation for the procedure
  * Inability to understand a Numeric Pain rating Scale due to cognitive dysfunction or linguistic barrier
  * Movement disorder making a person unable to lie still for the duration of the evaluation period.
  * Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper extremity complex regional pain syndrome treated at the pain clinic of the Maisonneuve-Rosemont Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Change in NoL index from baseline | 20 minutes
  • Change in the NoL index after a painful physiotherapy exercise in patients with upper limb CRPS 20 minutes after a stellate ganglion block, from baseline (before the stellate ganglion block)

SECONDARY OUTCOMES:
Change in peak NoL index values before and after a stellate ganglion block | 20 minutes
  Measure the change in peak NoL index (peak NoL index after a painful physiotherapy exercise before the stellate ganglion block minus the peak NoL index value after a painful physiotherapy exercise after the stellate ganglion block
change in Numeric Rating Scale (NRS) pain intensity score (from 0-10) before and after a stellate ganglion block | 20 minutes
  Measure the change in NRS pain intensity score after a painful physiotherapy exercise, before and 20 minutes after a stellate ganglion block.
correlation between change in NoL index and change in the Numeric Rating Scale (NRS) pain score (from 0-10) from baseline | 20 minutes
  Correlate the NoL index variation (delta NoL) with the NRS pain score variation (delta NRS) painful physiotherapy exercise in patients with upper limb CRPS, before and 20 minutes after a stellate ganglion block.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Brulotte, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No